CLINICAL TRIAL: NCT06112509
Title: Evolution of Vestibular Function After Treatment of a Vestibular Schwannoma by Gamma-knife
Brief Title: Evolution of Vestibular Function After Treatment of a Vestibular Schwannoma by Gamma-knife Radio-surgery
Acronym: EVERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/823
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vestibular Schwannoma; Neurinoma, Acoustic; Acoustic Neuroma
Keywords: vestibular; schwannoma; radiosurgery; gamma-knife; neurinoma; acoustic
MeSH Terms: conditions — Neuroma, Acoustic; Neurilemmoma

STUDY DESIGN:
Intervention Model Description: Prognostic cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiosurgery (Other)
  Interventions: Other: Vestibular exam

INTERVENTIONS:
Other: Vestibular exam — Interrogation, videonystagmoscopy, videonystagmography, video-head-impulse-test

SUMMARY:
The purpose of this study is to evaluate the vestibular effects of gamma-knife radiosurgery, as part of the treatment of vestibular schwannoma.

DETAILED DESCRIPTION:
Vestibular schwannoma is a benign tumor located on the vestibulocochlear nerve. It represents 6 to 8% of intracranial tumors, 80% of ponto-cerebral angle tumors and its frequency is 13 cases per million inhabitants per year.

The main symptoms related to the development of vestibular schwannoma are unilateral deafness of perception, unilateral tinnitus, unilateral vestibular deficit vertigo, facial paralysis.

Management is divided into 3 options: monitoring, surgery and gamma-knife radiosurgery.

This study will focus on gamma-knife radiosurgery. The objective of this treatment is to stabilize the evolution of schwannoma.

This study aims to describe the vestibular effects of radiosurgery.

ELIGIBILITY:
Inclusion Criteria :

* Men and women aged 18 to 90 included
* Subject who benefited from gamma-knife radiosurgery as part of the treatment of vestibular schwannoma
* Non-opposition of the subject to participate in the study
* Affiliation to a French social security scheme or beneficiary of such a scheme

Exclusion Criteria :

* Subject with another vestibular pathology
* Subject who did not benefit from a vestibular assessment before treatment with gamma-knife radiosurgery
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and/or weak cooperation anticipated by the investigator
* Subject without health insurance
* Subject being in the period of exclusion from another study or provided for by the "national volunteer file".

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Description of vestibular function with videonystagmography before gamma-knife radiosurgery, as part of the treatment of vestibular schwannoma. | 1 month before gamma-knife radiosurgery
  Videonystagmography: Results of caloric tests = Intervestibular deficit (in percentage)
Description of vestibular function with vidéonystagmoscopy before gamma-knife radiosurgery, as part of the treatment of vestibular schwannoma. | After gamma-knife radiosurgery at 6 month or 12 month or 18 month or 2 years or 3 years depending on the history of the treatment
  Videonystagmography: Results of caloric tests = Intervestibular deficit (in percentage)

SECONDARY OUTCOMES:
Description of vestibular symptoms before gamma-knife radiosurgery as part of the treatment of vestibular schwannoma. | 1 month before gamma-knife radiosurgery
  Dizziness Handicap Inventoryquestionnaire (DHI questionnaire)
Description of vestibular symptoms after gamma-knife radiosurgery as part of the treatment of vestibular schwannoma. | After gamma-knife radiosurgery at 6 month or 12 month or 18 month or 2 years or 3 years depending on the history of the treatment
  Dizziness Handicap Inventoryquestionnaire (DHI questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: DAMON Veronique, MD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France